CLINICAL TRIAL: NCT06417723
Title: Effect of Maxillary Nerve Block for Septoplasty
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Adiyaman University Research Hospital (Other)
Responsible Party: Principal Investigator, Nezir Yılmaz, Associate Professor,MD, Adiyaman University Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ADYU-ANS-NY-04
Record Dates: First submitted 2024-05-11; First posted 2024-05-16 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-05

CONDITIONS: Post Operative Pain
Keywords: postoperative pain; maxillary nerve block; septoplasty
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: two groups designed from septoplasty patintes for study.
  1. only general anesthesia
  2. General anesthesia + maxillary nerve block
Who Masked: Participant, Investigator
Masking Description: for patients - closed envelope system for investigator - Maxillary nerve block performer will not participate pain and results assesment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Block group (Experimental): Bilateral maxillary nerve block was planned to be performed using 10 cc 0.25% bupivacaine via suprazigomatic approach after providing airway safety in the block group with general anaesthesia applications. The haemodynamic values (blood pressure arterial, peak heart rate, peripheral oxygen saturation), postoperative numeric pain scores and postoperative quality of recovery index (QoR-15) values at the 24th hour will be recorded .
  Interventions: Procedure: Maxillary nerve block
- Control group (No Intervention): No intevention was planned for this group. Only genaeral anesthesia applications will use for surgery. The haemodynamic values (blood pressure arterial, peak heart rate, peripheral oxygen saturation), postoperative numeric pain scores and postoperative quality of recovery index (QoR-15) values at the 24th hour will be recorded .

INTERVENTIONS:
Procedure: Maxillary nerve block — It is aimed to reach the maxillary nerve trace with a peripheral nerve block needle using the suprazigomatic approach and to create a temporary block in the maxillary nerve with local anaesthetic injection.
  Arms: Block group

SUMMARY:
The aim of this study was to determine the effect of maxillary nerve blockage on both postoperative pain scores and recovery quality index in septoplasty operations. Thus, it was aimed to determine an alternative method that can be used in postoperative analgesia that will suppress postoperative pain complaints and increase the comfort level of patients after septoplasty operations.

DETAILED DESCRIPTION:
Patients who were planned to be operated for septoplasty at Adıyaman University Training and Research Hospital, who were informed about the study and agreed to participate in the study with their written consent were included in the study.

The patients who agreed to participate in the study were divided into two groups by closed envelope method and bilateral maxillary nerve blockade was planned to be performed using 10 cc 0.25% bupivacaine via suprazigomatic approach after providing airway safety in the block group with general anaesthesia applications in both groups. The haemodynamic values (blood pressure arterial, peak heart rate, peripheral oxygen saturation), postoperative numeric pain scores and postoperative quality of recovery index (QoR-15) values at the 24th hour were recorded and these values were compared in both groups.

Thus, it was aimed to evaluate the effects of maxillary nerve blockade in septoplasty operations.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II , Septoplasty patints

Exclusion Criteria:

* ASA III-IV
* Deny to participte in study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-09-15 (Estimated)

PRIMARY OUTCOMES:
The visual analog pain score | three months
  The visual analog scale (VAS) is a validated, subjective measure for acute and chronic pain. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" and "worst pain."

SECONDARY OUTCOMES:
Quality of recovery (QoR -15) | three months
  The QoR-15 scale is a unidimensional measurement of quality of recovery measured in five domains: physical comfort, pain, physical independence, psychological support, and emotional state. The QoR-15 scale provides a score ranging from 0 to 150, with a high score indicating a good quality of recovery

CONTACTS AND LOCATIONS:
Locations (1):
- Adıyaman Training and Research Hospital, Adıyaman, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided